CLINICAL TRIAL: NCT02336997
Title: Evaluation of the Effect of Autologous Fat and SVF Transplantation in Promoting Mechanical-stretch Induced in Vivo Skin Regeneration
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qing-FengLi Li,MD (Other)
Responsible Party: Sponsor-Investigator, Qing-FengLi Li,MD, Prof., Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: [2014]47
Record Dates: First submitted 2014-12-26; First posted 2015-01-13 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Scar
Keywords: skin regeneration; mechanical stretch
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- FAT-GRAFT (Experimental): Fat graft transplantation
  Interventions: Procedure: FAT-GRAFT
- SVF-TRANSPLANTATION (Experimental): Transplantation of resuspended SVF
  Interventions: Procedure: SVF-TRANSPLANTATION
- CONTROL (Placebo Comparator): Same volume saline injection
  Interventions: Procedure: PLACEBO

INTERVENTIONS:
Procedure: FAT-GRAFT — Liposuction will be performed and autologous fat graft will be harvest after washing with saline. Patients will receive autologous fat graft transplantation subdermally to expanded skin at the density of 0.1 ml/cm2.
  Arms: FAT-GRAFT
Procedure: SVF-TRANSPLANTATION — Liposuction will be performed. SVF will be separated from autologous fat graft by collagenase digestion. Patients will receive resuspended SVF transplantation subdermally to expanded skin at the density of 1*10e6 cells/cm2.
  Arms: SVF-TRANSPLANTATION
Procedure: PLACEBO — Saline will be injected into expanded skin.
  Arms: CONTROL

SUMMARY:
The purpose of this study is to evaluating whether autologous grafted fat transplantation or SVF transplantation is safe and/or effective to accelerating skin regeneration and soft tissue expansion.

DETAILED DESCRIPTION:
Reconstruction of large scale skin defect is a challenge to clinical surgeons. Soft tissue expansion has won wide attention in recent years as it promotes skin regeneration with perfectly matched tissue. However, some patients with poor skin regenerative ability would suffer from skin flap over-thinned and even necrosis under the continuous stretching by silicone expander. This study is to evaluate the effects of autologous fat graft/SVF transplantation on accelerating skin regeneration and promoting tissue expansion process.

Patients aged between 18 to 60 years old who appear with deteriorated expanded skin will be enrolled and randomized into three groups, named as the experimental group and the control group. Patients from the FAT-GRAFT group will have a liposuction and subdermal fat graft transplantation. Patients from the SVF-TRANSPLANTATION group will have a liposuction and SVF will be separated and transplanted intradermally to expanded skin. Patients from the control group will have saline injection.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Age of 18 to 60 years;
* Expanding skin donor site at the face, neck, anterior chest wall, abdominal wall or back;
* Implanted silicone expander of 80 to 600 ml in size;
* History of deterioration in the expanded skin texture that did not improve after the inflation procedure was suspended for more than 2 weeks;
* Persistent high level of expander internal pressure;
* Need for further skin expansion;

Exclusion Criteria:

* Not fit for soft tissue expansion treatment;
* Evidence of infection, ischemia, ulcer or other pathological changes within the targeting area which defined as not suitable for expansion; or history of delayed healing, radiational therapy;
* Significant renal, cardiovascular, hepatic and psychiatric diseases;
* Significant medical diseases or infection (including but not limited to the carrier of hepatitis B virus or HIV)
* BMI >30;
* History of any hematological disease, including leukopenia , thrombocytopenia, or thrombocytosis;
* History of allogenic bone marrow transplantation;
* Long history of smoking;
* Evidence of malignant diseases or unwillingness to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Occurence of Major Adverse Events | Up to approximately 24 months after study start
  Including expanded flap ischaemia, necrosis, fluidify, infection, and all other adverse events
To Measure the Change in Inflation Volume of the Silicone Expander from Baseline at 8 weeks | baseline and 8 weeks post treatment
  Record the inflation volume of each expander with the maintained inner pressure.

SECONDARY OUTCOMES:
To Measure the Size of Expanded Flap with 3D laser scanner and calculate the surface of expanded skin | baseline and 8 weeks post treatment
  Record the outface of expanded skin flap with 3D laser scanner and calculate the surface of expanded skin
To Measure the Texture of Expanded Flap with VISIA scanner | 4 weeks and 8 weeks post treatment
  Evaluate skin texture with VISIA scanner and compare the characteristics
To Measure Expanded Skin Thickness by Ultrasound Scanning | baseline, 4 weeks and 8 weeks post treatment
  Measure the dermal and epidermal thickness of expanded skin by ultrasound scanning

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Ninth People's Hospital, Affliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai